CLINICAL TRIAL: NCT03032263
Title: A Comparison of Direct Laryngoscopy and Video Laryngoscopy Using the C-Mac in Pediatric Nasal Intubations
Brief Title: Video vs. Direct Laryngoscopy in Pediatric Nasal Intubation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMac-032016
Record Dates: First submitted 2017-01-12; First posted 2017-01-26 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Nasal Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Laryngoscopy (Active Comparator): These patients will be nasally intubated for their procedure via direct laryngoscopy. We will observe and record incidence of Magill forcep use, presence or absence of nasal bleeding, and the grade of laryngeal view. We will also record any general narrative comments from the provider about the ease or difficulty of intubation.
  Interventions: Device: Direct Laryngoscopy
- Video Laryngoscopy (Experimental): These patients will undergo Video Laryngoscopy for nasal intubation. We will observe and record incidence of Magill forcep use, presence or absence of nasal bleeding, and the grade of laryngeal view. We will also record any general narrative comments from the provider about the ease or difficulty of intubation.
  Interventions: Device: Video Laryngoscopy for nasal intubation

INTERVENTIONS:
Device: Video Laryngoscopy for nasal intubation — The anesthesia provider will use a video laryngoscope to facilitate the nasal intubation for the procedure.
  Arms: Video Laryngoscopy
Device: Direct Laryngoscopy — These patients will be nasally intubated for their procedure via direct laryngoscopy
  Arms: Direct Laryngoscopy

SUMMARY:
Nasal intubation is frequently used for dental procedures to promote an unimpeded view of the oral cavity. A nasal RAE endotracheal tube is longer than a standard oral endotracheal tube (ETT) and it is shaped so that end of the tube which attaches to the ventilator exits upward toward the forehead. This unique shape ensures that the tube will not interfere with surgical exposure of the oral cavity and mandible. The nasal RAE ETT can be placed in the trachea using either direct laryngoscopy (DL) or video laryngoscopy (C-Mac) . Sometimes this is possible without an adjuvant, but frequently a pair of specially shaped forceps, known as Magill forceps, is required to guide the distal tip of the Nasal RAE into the glottis due to the curvature of these ETT. Magill forceps are introduced into the mouth and are used to grasp the distal end of the Nasal RAE and direct it into the glottis. Contrary to what the current literature suggests, it has been our experience that nasal intubations using the C-Mac frequently do not require the use of Magill forceps at nearly the same rate as DL. This technique may improve the time and ease to intubation because of not having to use the Magill forceps. The use of Magill forceps can be awkward for the clinician, with poor visualization due to obstruction of the view by this tool in the airway, and small working space within the posterior oropharynx. For these reasons, the possibility of not having to use Magill forceps because the investigators are using a C-Mac as the only tool to intubate is a potentially inviting one.

DETAILED DESCRIPTION:
The objective of this study is to compare the need for the use of standard Magill forceps when performing a nasal intubation with either conventional DL or VL with a C-Mac. Secondarily the investigators will also examine the time to intubate (TTI) for both methods as well.

Once the patient is recruited, the patient will then be randomized to either intubation using DL or VL with a C-Mac. Once the patient is under anesthesia, the intubation will be performed by an attending pediatric anesthesiologist or experience pediatric CRNA who has experience both DL and with the C-Mac and will attempt to intubate the patient with or without Magill forceps as needed.

The investigators will record the time to intubation (TTI) from the time the laryngoscope or C-Mac is placed in the mouth to the first appearance of end tidal carbon dioxide (ETCO2). the investigators will record the presence or absence of nasal bleeding, and the grade of laryngeal view. The investigators will also record any general narrative comments about the ease or difficulty of intubation in both groups.

The study will be performed at Wake Forest Baptist Medical Center.

Patients between the ages of 3 and 14 scheduled for comprehensive dental treatment under general anesthesia will be included.

Normal appearing airway upon pre-operative assessment. The investigators have calculated a sample size of 35 patients in each group to be able to detect a significant difference in the rate of use of Magill forceps to place a nasal RAE ETT in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 3 and 14 scheduled for comprehensive dental treatment under general anesthesia
* Normal appearing airway upon pre-operative assessment

Exclusion Criteria:

* Patient with a history of difficult airway/intubation
* Patients suspected to have a difficult airway
* History of cleft palate and/or cleft palate repair
* Pregnancy
* Emergency status of surgery
* Any patient with a contra-indication to nasal tube placement
* Any patient with a potentially increased risk of nasal bleeding from nasal placement of the ETT i.e. patients on aspirin or other anticoagulants, patient's with hemophilia

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Lu Y, Huang Y, Jiang H. Pediatric video laryngoscope versus direct laryngoscope: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2014 Oct;24(10):1056-65. doi: 10.1111/pan.12458. Epub 2014 Jun 24. PMID 24958249
- [Result] Kim HJ, Kim JT, Kim HS, Kim CS, Kim SD. A comparison of GlideScope((R)) videolaryngoscopy and direct laryngoscopy for nasotracheal intubation in children. Paediatr Anaesth. 2011 Apr;21(4):417-21. doi: 10.1111/j.1460-9592.2010.03517.x. Epub 2011 Jan 19. PMID 21244568
- [Result] Jones PM, Armstrong KP, Armstrong PM, Cherry RA, Harle CC, Hoogstra J, Turkstra TP. A comparison of glidescope videolaryngoscopy to direct laryngoscopy for nasotracheal intubation. Anesth Analg. 2008 Jul;107(1):144-8. doi: 10.1213/ane.0b013e31816d15c9. PMID 18635480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.33 (2.16) | 7.33 (4.55) | 6.83 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Use of Magill Forceps for Nasal Intubations
Description: Reported as the number and percentage of participants that needed the use of Magill forceps during intubation
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 6 | 6
Participants | 1 | 2

2. Secondary Outcome: Time to Intubation
Description: Reported as the average time it took to intubate (seconds).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 6 | 6
seconds | 68.43 (81.1) | 57.1 (25.12)

3. Secondary Outcome: Grade of Larynx View
Description: Larynx view is graded from 1-4 (1 is full glottis visible, 2 is only posterior commisure, 3 is only epiglottis visible, and 4 is no glottis structures are visible).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 6 | 6
units on a scale | 1.33 (.52) | 1 (0)

4. Secondary Outcome: Presence of Nasal Bleeding
Description: Number of participants that experienced nasal bleeding was recorded.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 6 | 6
Participants | 3 | 3

5. Secondary Outcome: Incidence of Failed Nasal Intubation
Description: The incidence of failed nasal intubation was recorded as the number of intubations that were not successful.
Time Frame: 1 day
Measure: Number; unit: number of intubations
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
Number analyzed (Participants) | 6 | 6
number of intubations | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Direct Laryngoscopy | Video Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT03032263/Prot_SAP_001.pdf